CLINICAL TRIAL: NCT01872702
Title: Targeted Chemo-elimination (TCE) to Eradicate Malaria in Areas of Suspected or Proven Artemisinin Resistance in Southeast Asia and South Asia
Brief Title: Targeted Chemo-elimination (TCE) of Malaria
Acronym: TME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Mahidol Oxford Tropical Medicine Research Unit (Other); National Centre for Parasitology, Entomology and Malaria Control, Cambodia (Other); FHI 360 (Other); Oxford University Clinical Research Unit, Vietnam (Other); National Malaria Control Program, Vietnam (Other Government); Myanmar Oxford Clinical Research Unit (Other); National Malaria Control Program, Myanmar (Other Government); Lao-Oxford-Mahosot Hospital Wellcome Trust Research Unit (Other); Shoklo Malaria Research Unit (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BAKMAL1305
Record Dates: First submitted 2013-06-04; First posted 2013-06-07 (Estimated); Last update posted 2020-08-28 (Actual); Status verified 2017-08

CONDITIONS: Plasmodium Falciparum Malaria
Keywords: Malaria elimination; Chemotherapy; Epidemiology; South East Asia; Artemisinin resistance; Dihydroartemisinin piperaquine; Primaquine
MeSH Terms: conditions — Malaria, Falciparum | interventions — Primaquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- malaria elimination using DP and low-dose primaquine (Experimental): Two villages randomly allocated to intervention (chemo-elimination) at each of the 4 sites (population approximately 500 people in each village). In these villages the entire population will be invited to receive three, monthly rounds of treatment with dihydroartemisinin-piperaquine and primaqunine to kill malaria parasites. The micro-epidemiology of malaria will be studied and prevalence and patterns of transmission used for comparison. NB, in Cambodia there will be no intervention villages and all four villages will be used to study the micro-epidemiology of malaria transmission in the absence of malaria elimination.
  Interventions: Drug: malaria elimination using DP and low-dose primaquine
- Control villages (No Intervention): Two villages randomly allocated to control (no chemo-elimination) at each of the 4 sites (population approximately 500 people in each village). In these villages only the micro-epidemiology of malaria will be studied and prevalence and patterns of transmission used for comparison. NB, in Cambodia there will be no intervention villages and all four villages will be used to study the micro-epidemiology of malaria transmission in the absence of malaria elimination.
  From June 2013 to June 2014 Cambodia site conducted surveys with no medical intervention (treatment arm). In July 2015 Cambodia implemented the TCE protocol with two intervention and two control villages. Primaquine is not used in the TCE treatment regimen in Cambodia. Both studies were approved under OxTREC reference no. 1017-13 and 1015-13.

INTERVENTIONS:
Drug: malaria elimination using DP and low-dose primaquine — Treatment of all persons resident in the intervention villages including those who do not have malaria parasites as detected by rapid diagnostic test. This is to interrupt p.f malaria transmission by removing the reservoir of all potentially infectious people from the area.
  Other Names: Three monthly rounds of:; Dihydroartemisinin-piperaquine; Low-dose primaquine
  Arms: malaria elimination using DP and low-dose primaquine

SUMMARY:
The overall aim of this study is two fold:

1. to pilot targeted chemo-elimination of plasmodium falciparum malaria in known areas of artemisinin resistance in South East Asia.
2. to understand the micro-epidemiology of malaria in these areas; chiefly, the prevalence and importance to on-going transmission of sub-clinical p.f malaria infections.

DETAILED DESCRIPTION:
The spread of artemisinin resistance in Plasmodium falciparum, which compromises the therapeutic efficacy of artemisinin combination treatments (ACTs), is the greatest threat to current global initiatives to control and eliminate malaria and is considered the highest priority of the WHO Global Malaria Programme. If not eliminated, resistant parasites could spread across Asia to Africa, as happened with resistance to other antimalarials in the past.

Conventional descriptions of the epidemiology of malaria in low transmission settings suggest that malaria prevalences are low (<10%) and heterogeneous. Most or all infections are thought to be symptomatic so the focus of malaria control activities is on the identification and treatment of symptomatic individuals. We and others have shown recently that artemisinin resistant P. falciparum is prevalent in Western Cambodia, and that it is now also found along the Thailand-Myanmar border and Vietnam. We have recently developed highly sensitive quantitative PCR (uPCR) methods for parasite detection using >1mL of blood which are 5,000 times more sensitive than conventional microscopy, and 100 times more sensitive than currently used PCR.

We have studied villages along the Thai-Myanmar border which are typical for the region and are classified by conventional epidemiological techniques as low-transmission (5-20% malaria prevalence). Our studies suggest that the majority of the population is infected. In Pailin, Western Cambodia, in areas where the National Malaria Control Programme and WHO believe that malaria has been all but eliminated, we have also found very high rates (>80%) of sub-microscopic parasitaemia in patients with fever or history of fever who are RDT negative. Thus, there is a lot more asymptomatic malaria in low transmission settings than previously thought, suggesting that control and elimination activities need to be rethought.

Highly sensitive quantitative PCR (uPCR) requires a venous blood sample, a laboratory which can perform vacuum DNA extraction, and on average four weeks for processing. A rapid highly sensitive diagnostic test which can be performed at the point of care would be a technological breakthrough. Screening with highly sensitive RDTs and treating of asymptomatic carriers will have a range of public health applications. Such tests are becoming available in 2017 and will be evaluated side by side with uPCR.

This study is designed to conduct and evaluate the efficacy of pilot implementation of targeted chemo-elimination in selected areas with the goal of eliminating malaria in these regions. This differs from mass drug administration (MDA); it is a strategy used to identify specific areas where mass treatment is necessary, in this case to eliminate all malaria parasites. Elimination will be targeted at communities with significant levels of subclinical infection and transmission which will be identifiable in the future by comparing rates of positivity by RDT or microscopy from new population samples against our qPCR data, which shows the true falciparum prevalence.

The study will assess the feasibility, safety and acceptability of this strategy and its impact on the transmission of malaria and the progression of artemisinin resistance. In addition it will evaluate the contribution of low parasitaemia carriage to transmission of artemisinin resistant malaria. These pilot studies are a necessary prelude to future scale up and policy implementation.

Dihydroartemisinin-piperaquine (DP) is a highly efficacious and inexpensive ACT which is well tolerated by all age groups when used to treat uncomplicated multi-drug resistant falciparum malaria in South East Asia. Monthly DP treatments have proved highly effective and well tolerated. When used as part of a MDA strategy, the addition of a gametocytocidal drug contributes towards the goal of malaria elimination by adding a strong transmission blocking activity to the regimen. Primaquine (PQ), the only currently licensed 8-aminoquinoline, is relatively safe and very effective when used at a dose of 0.25 mg base/kg, and does not require G6PD screening. Thus, we propose to evaluate the potential of this strategy to eliminatie malaria focally in areas where artemisinin resistance in P. falciparum is prevalent using DP plus PQ.

ELIGIBILITY:
OxTREC reference: 1017-13

Inclusion Criteria:

* Age ≥6 months, male or female,
* Written informed consent (by parent/guardian in case of children)

Exclusion Criteria:

* Pregnant women will not receive primaquine (urine pregnancy tests will be performed on women of appropriate age groups before drug administration at each TCE round)
* History of allergy or known contraindication to artemisinins, piperaquine or PQ
* Those who are, in the opinion of the study clinician, ill at the time of drug administration

OxTREC reference: 1015-13

Inclusion Criteria

* Age ≥6 months, male or female,
* Written informed consent (by legally acceptable representative in case of children)
* Healthy at the time of the survey or drug administration
* Not pregnant

Exclusion Criteria

* Significant non-compliance with study requirements
* Loss to follow up
* Suspected severe adverse events
* Severe illness

OxTREC reference: 23-15

Part 1. qPCR survey for identification of potential TMT villages;

Inclusion criteria:

* Males and females 18 and above
* Written informed consent

Exclusion criteria:

* Pregnant women in their first trimester
* Presence of any acute severe illness at the time of survey

Part 2. TMT villages will be given directly observed therapy (DOT) with DP for 3 days and PQ (0.25 mg/kg) will be given on day 1

Inclusion criteria for TMT

* Age ≥one year, male and female,
* Willing to provide consent for those 18 years and above. For children 10-18 years old, parents/guardians must provide consent, and the children must provide assent. For children below 10 years old, the parents/guardians must provide consent.

Exclusion criteria for TMT

* History of allergy or known contraindication to artemisinins, piperaquine or PQ.
* Refusal of treatment.
* Pregnant women in their 1st trimester.

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 8000 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
prevalence of falciparum malaria measured by qPCR (quantitative real time polymerase chain reaction), 12 months after the first administration of treatment with dihydroartemisinin-piperaquine and primaquine. (1017-13 and 23-15) | 12 months
  Percentage falls in asymptomatic malaria prevalence in the intervention villages vs control villages, as determined by highly sensitive qPCR, 12 months after the first administration of treatment with dihydroartemisinin-piperaquine and primaquine.
prevalence of falciparum malaria measured by qPCR (quantitative real time polymerase chain reaction), 12 months after the first administration of targeted malaria elimination (1015-13) | 12 months
  Percentage falls in asymptomatic malaria prevalence in the intervention villages vs control villages, as determined by highly sensitive qPCR, 12 months after the first administration of treatment with dihydroartemisinin-piperaquine
prevalence of falciparum malaria measured by qPCR (quantitative real time polymerase chain reaction), 4 months after the first administration of target malaria-elimination (23-15) | 4 months
  Percentage falls in asymptomatic malaria prevalence in the intervention villages vs control villages, as determined by highly sensitive qPCR, 4 months after the first administration of treatment with dihydroartemisinin-piperaquine and primaquine.

SECONDARY OUTCOMES:
Safety and acceptability of targeted malaria elimination (1017-13 and 1015-13) | 12 months
  Safety and acceptability of targeted malaria elimination, evaluated by questionnaires filled out by participants or care givers.

OTHER OUTCOMES:
Effect on gametocyte carriage by targeted malaria elimination (1017-13 and 1015-13) | 12 months
  Effect on gametocyte carriage by targeted malaria elimination, measured by the proportions of gametocyte carriers over the 12 month period
Characterize parasite carriage using highly sensitive techniques in four geographically separate sites where resistance to artemisinin has been documented (1017-13 and 1015-13) | 12 months
  Characterize parasite carriage using by molecular analysis of parasite genotypes, markers of resistance and parasite population genetic structure
Acceptability of targeted Chemo-elimination of malaria measured by number of peaople participate (1017-13) | 12 months
Cost estimates of targeted Chemo-elimination of malaria by sampling strategy (1017-13) | 12 months
incidence of clinical malaria in the villages over the first 12 months (1015-13) | 12 months
The proportion of Artemisinin resistance - P.falciparum infections (23-15) | 12 months
Sensitivity of novel RDTs (HS RDT) | 12 months
  (Laos site only)
Specificity of novel RDTs (HS RDT) | 12 months
  (Laos site only)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas J White, PhD, Principal Investigator — University of Oxford
Locations (5):
- Mahidol Oxford Clincal Research Unit, Myanmar, Rangoon, Burma
- Pailin, Pailin, Cambodia
- Savannakhet, Savannakhet, Laos
- Shoklo Malaria Research Unit, Mae Sot, Changwat Tak, Thailand
- Oxford University Clinical Research Unit - Vietnam, Ho Chi Minh City, Vietnam

REFERENCES:
- [Background] (2011) Global Plan for Artemisinin Resistance Containment. Geneva: World Health Organisation.
- [Background] Dondorp AM, Nosten F, Yi P, Das D, Phyo AP, Tarning J, Lwin KM, Ariey F, Hanpithakpong W, Lee SJ, Ringwald P, Silamut K, Imwong M, Chotivanich K, Lim P, Herdman T, An SS, Yeung S, Singhasivanon P, Day NP, Lindegardh N, Socheat D, White NJ. Artemisinin resistance in Plasmodium falciparum malaria. N Engl J Med. 2009 Jul 30;361(5):455-67. doi: 10.1056/NEJMoa0808859. PMID 19641202
- [Background] Phyo AP, Nkhoma S, Stepniewska K, Ashley EA, Nair S, McGready R, ler Moo C, Al-Saai S, Dondorp AM, Lwin KM, Singhasivanon P, Day NP, White NJ, Anderson TJ, Nosten F. Emergence of artemisinin-resistant malaria on the western border of Thailand: a longitudinal study. Lancet. 2012 May 26;379(9830):1960-6. doi: 10.1016/S0140-6736(12)60484-X. Epub 2012 Apr 5. PMID 22484134
- [Background] Hien TT, Thuy-Nhien NT, Phu NH, Boni MF, Thanh NV, Nha-Ca NT, Thai le H, Thai CQ, Toi PV, Thuan PD, Long le T, Dong le T, Merson L, Dolecek C, Stepniewska K, Ringwald P, White NJ, Farrar J, Wolbers M. In vivo susceptibility of Plasmodium falciparum to artesunate in Binh Phuoc Province, Vietnam. Malar J. 2012 Oct 26;11:355. doi: 10.1186/1475-2875-11-355. PMID 23101492
- [Background] Amaratunga C, Sreng S, Suon S, Phelps ES, Stepniewska K, Lim P, Zhou C, Mao S, Anderson JM, Lindegardh N, Jiang H, Song J, Su XZ, White NJ, Dondorp AM, Anderson TJ, Fay MP, Mu J, Duong S, Fairhurst RM. Artemisinin-resistant Plasmodium falciparum in Pursat province, western Cambodia: a parasite clearance rate study. Lancet Infect Dis. 2012 Nov;12(11):851-8. doi: 10.1016/S1473-3099(12)70181-0. Epub 2012 Aug 30. PMID 22940027
- [Background] Tran TH, Dolecek C, Pham PM, Nguyen TD, Nguyen TT, Le HT, Dong TH, Tran TT, Stepniewska K, White NJ, Farrar J. Dihydroartemisinin-piperaquine against multidrug-resistant Plasmodium falciparum malaria in Vietnam: randomised clinical trial. Lancet. 2004 Jan 3;363(9402):18-22. doi: 10.1016/s0140-6736(03)15163-x. PMID 14723988
- [Background] Smithuis F, Kyaw MK, Phe O, Aye KZ, Htet L, Barends M, Lindegardh N, Singtoroj T, Ashley E, Lwin S, Stepniewska K, White NJ. Efficacy and effectiveness of dihydroartemisinin-piperaquine versus artesunate-mefloquine in falciparum malaria: an open-label randomised comparison. Lancet. 2006 Jun 24;367(9528):2075-85. doi: 10.1016/S0140-6736(06)68931-9. PMID 16798391
- [Background] Ashley EA, Krudsood S, Phaiphun L, Srivilairit S, McGready R, Leowattana W, Hutagalung R, Wilairatana P, Brockman A, Looareesuwan S, Nosten F, White NJ. Randomized, controlled dose-optimization studies of dihydroartemisinin-piperaquine for the treatment of uncomplicated multidrug-resistant falciparum malaria in Thailand. J Infect Dis. 2004 Nov 15;190(10):1773-82. doi: 10.1086/425015. Epub 2004 Oct 18. PMID 15499533
- [Background] Ashley EA, McGready R, Hutagalung R, Phaiphun L, Slight T, Proux S, Thwai KL, Barends M, Looareesuwan S, White NJ, Nosten F. A randomized, controlled study of a simple, once-daily regimen of dihydroartemisinin-piperaquine for the treatment of uncomplicated, multidrug-resistant falciparum malaria. Clin Infect Dis. 2005 Aug 15;41(4):425-32. doi: 10.1086/432011. Epub 2005 Jul 15. PMID 16028147
- [Background] White NJ, Qiao LG, Qi G, Luzzatto L. Rationale for recommending a lower dose of primaquine as a Plasmodium falciparum gametocytocide in populations where G6PD deficiency is common. Malar J. 2012 Dec 14;11:418. doi: 10.1186/1475-2875-11-418. PMID 23237606
- [Background] Myint HY, Ashley EA, Day NP, Nosten F, White NJ. Efficacy and safety of dihydroartemisinin-piperaquine. Trans R Soc Trop Med Hyg. 2007 Sep;101(9):858-66. doi: 10.1016/j.trstmh.2007.05.018. Epub 2007 Jul 19. PMID 17659311
- [Derived] Shah MP, Hwang J, Choi L, Lindblade KA, Kachur SP, Desai M. Mass drug administration for malaria. Cochrane Database Syst Rev. 2021 Sep 29;9(9):CD008846. doi: 10.1002/14651858.CD008846.pub3. PMID 34585740
- [Derived] McLean ARD, Indrasuta C, Khant ZS, Phyo AK, Maung SM, Heaton J, Aung H, Aung Y, Soe K, Swe MMM, von Seidlein L, Tun NN, Tun KM, Day NPJ, Ashley EA, Hlaing T, Kyaw TT, Dondorp AM, Imwong M, White NJ, Smithuis FM. Mass drug administration for the acceleration of malaria elimination in a region of Myanmar with artemisinin-resistant falciparum malaria: a cluster-randomised trial. Lancet Infect Dis. 2021 Nov;21(11):1579-1589. doi: 10.1016/S1473-3099(20)30997-X. Epub 2021 Jun 18. PMID 34147154
- [Derived] von Seidlein L, Peerawaranun P, Mukaka M, Nosten FH, Nguyen TN, Hien TT, Tripura R, Peto TJ, Pongvongsa T, Phommasone K, Mayxay M, Imwong M, Watson J, Pukrittayakamee S, Day NPJ, Dondorp AM. The probability of a sequential Plasmodium vivax infection following asymptomatic Plasmodium falciparum and P. vivax infections in Myanmar, Vietnam, Cambodia, and Laos. Malar J. 2019 Dec 30;18(1):449. doi: 10.1186/s12936-019-3087-1. PMID 31888643
- [Derived] Peerawaranun P, Landier J, Nosten FH, Nguyen TN, Hien TT, Tripura R, Peto TJ, Phommasone K, Mayxay M, Day NPJ, Dondorp A, White N, von Seidlein L, Mukaka M. Intracluster correlation coefficients in the Greater Mekong Subregion for sample size calculations of cluster randomized malaria trials. Malar J. 2019 Dec 18;18(1):428. doi: 10.1186/s12936-019-3062-x. PMID 31852499
- [Derived] von Seidlein L, Peto TJ, Landier J, Nguyen TN, Tripura R, Phommasone K, Pongvongsa T, Lwin KM, Keereecharoen L, Kajeechiwa L, Thwin MM, Parker DM, Wiladphaingern J, Nosten S, Proux S, Corbel V, Tuong-Vy N, Phuc-Nhi TL, Son DH, Huong-Thu PN, Tuyen NTK, Tien NT, Dong LT, Hue DV, Quang HH, Nguon C, Davoeung C, Rekol H, Adhikari B, Henriques G, Phongmany P, Suangkanarat P, Jeeyapant A, Vihokhern B, van der Pluijm RW, Lubell Y, White LJ, Aguas R, Promnarate C, Sirithiranont P, Malleret B, Renia L, Onsjo C, Chan XH, Chalk J, Miotto O, Patumrat K, Chotivanich K, Hanboonkunupakarn B, Jittmala P, Kaehler N, Cheah PY, Pell C, Dhorda M, Imwong M, Snounou G, Mukaka M, Peerawaranun P, Lee SJ, Simpson JA, Pukrittayakamee S, Singhasivanon P, Grobusch MP, Cobelens F, Smithuis F, Newton PN, Thwaites GE, Day NPJ, Mayxay M, Hien TT, Nosten FH, Dondorp AM, White NJ. The impact of targeted malaria elimination with mass drug administrations on falciparum malaria in Southeast Asia: A cluster randomised trial. PLoS Med. 2019 Feb 15;16(2):e1002745. doi: 10.1371/journal.pmed.1002745. eCollection 2019 Feb. PMID 30768615
- [Derived] Pongvongsa T, Phommasone K, Adhikari B, Henriques G, Chotivanich K, Hanboonkunupakarn B, Mukaka M, Peerawaranun P, von Seidlein L, Day NPJ, White NJ, Dondorp AM, Imwong M, Newton PN, Singhasivanon P, Mayxay M, Pukrittayakamee S. The dynamic of asymptomatic Plasmodium falciparum infections following mass drug administrations with dihydroarteminisin-piperaquine plus a single low dose of primaquine in Savannakhet Province, Laos. Malar J. 2018 Nov 3;17(1):405. doi: 10.1186/s12936-018-2541-9. PMID 30390647
- [Derived] Imwong M, Madmanee W, Suwannasin K, Kunasol C, Peto TJ, Tripura R, von Seidlein L, Nguon C, Davoeung C, Day NPJ, Dondorp AM, White NJ. Asymptomatic Natural Human Infections With the Simian Malaria Parasites Plasmodium cynomolgi and Plasmodium knowlesi. J Infect Dis. 2019 Feb 15;219(5):695-702. doi: 10.1093/infdis/jiy519. PMID 30295822
- [Derived] Henriques G, Phommasone K, Tripura R, Peto TJ, Raut S, Snethlage C, Sambo I, Sanann N, Nguon C, Adhikari B, Pongvongsa T, Imwong M, von Seidlein L, Day NP, White NJ, Dondorp AM, Newton P, Ley B, Mayxay M. Comparison of glucose-6 phosphate dehydrogenase status by fluorescent spot test and rapid diagnostic test in Lao PDR and Cambodia. Malar J. 2018 Jun 22;17(1):243. doi: 10.1186/s12936-018-2390-6. PMID 29929514
- [Derived] Peto TJ, Tripura R, Sanann N, Adhikari B, Callery J, Droogleever M, Heng C, Cheah PY, Davoeung C, Nguon C, von Seidlein L, Dondorp AM, Pell C. The feasibility and acceptability of mass drug administration for malaria in Cambodia: a mixed-methods study. Trans R Soc Trop Med Hyg. 2018 Jun 1;112(6):264-271. doi: 10.1093/trstmh/try053. PMID 29917147
- [Derived] Tripura R, Peto TJ, Chea N, Chan D, Mukaka M, Sirithiranont P, Dhorda M, Promnarate C, Imwong M, von Seidlein L, Duanguppama J, Patumrat K, Huy R, Grobusch MP, Day NPJ, White NJ, Dondorp AM. A Controlled Trial of Mass Drug Administration to Interrupt Transmission of Multidrug-Resistant Falciparum Malaria in Cambodian Villages. Clin Infect Dis. 2018 Aug 31;67(6):817-826. doi: 10.1093/cid/ciy196. PMID 29522113
- [Derived] Peto TJ, Tripura R, Davoeung C, Nguon C, Nou S, Heng C, Kunthea P, Adhikari B, Lim R, James N, Pell C, Cheah PY. Reflections on a Community Engagement Strategy for Mass Antimalarial Drug Administration in Cambodia. Am J Trop Med Hyg. 2018 Jan;98(1):100-104. doi: 10.4269/ajtmh.17-0428. PMID 29165227
- [Derived] Tripura R, Peto TJ, Veugen CC, Nguon C, Davoeung C, James N, Dhorda M, Maude RJ, Duanguppama J, Patumrat K, Imwong M, von Seidlein L, Grobusch MP, White NJ, Dondorp AM. Submicroscopic Plasmodium prevalence in relation to malaria incidence in 20 villages in western Cambodia. Malar J. 2017 Jan 31;16(1):56. doi: 10.1186/s12936-017-1703-5. PMID 28143518
- [Derived] Tripura R, Peto TJ, Chalk J, Lee SJ, Sirithiranont P, Nguon C, Dhorda M, von Seidlein L, Maude RJ, Day NP, Imwong M, White NJ, Dondorp AM. Persistent Plasmodium falciparum and Plasmodium vivax infections in a western Cambodian population: implications for prevention, treatment and elimination strategies. Malar J. 2016 Mar 24;15:181. doi: 10.1186/s12936-016-1224-7. PMID 27013512
- [Derived] Bancone G, Chowwiwat N, Somsakchaicharoen R, Poodpanya L, Moo PK, Gornsawun G, Kajeechiwa L, Thwin MM, Rakthinthong S, Nosten S, Thinraow S, Nyo SN, Ling CL, Wiladphaingern J, Kiricharoen NL, Moore KA, White NJ, Nosten F. Single Low Dose Primaquine (0.25 mg/kg) Does Not Cause Clinically Significant Haemolysis in G6PD Deficient Subjects. PLoS One. 2016 Mar 24;11(3):e0151898. doi: 10.1371/journal.pone.0151898. eCollection 2016. PMID 27010542
- See also: The Mahidol Oxford Tropical Medicine Research Unit — http://www.tropmedres.ac